CLINICAL TRIAL: NCT05459909
Title: A Study of the Effect of Synbiotic Supplementation and/or Dietary Intervention With Fruits and Vegetables on the Risk of Metabolic Dysfunction and Overweight or Obesity Among Hong Kong Chinese
Brief Title: The Effect of Synbiotic and Diet Modification Among Overweight or Obese Hong Kong Chinese
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lauw Susana, Principal Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYN-DIET-OB-RCT
Record Dates: First submitted 2022-07-07; First posted 2022-07-15 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Obesity
Keywords: Obesity; Overweight; Synbiotic; Diet; Metabolic dysfunction
MeSH Terms: conditions — Obesity; Overweight | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Synbiotic supplementation (Experimental): Synbiotic supplementation
  Interventions: Dietary Supplement: Synbiotic supplementation
- Dietary intervention (Experimental): Dietary intervention
  Interventions: Behavioral: Dietary intervention
- Synbiotic supplementation & dietary intervention (Experimental): Synbiotic supplementation & dietary intervention
  Interventions: Dietary Supplement: Synbiotic supplementation; Behavioral: Dietary intervention

INTERVENTIONS:
Dietary Supplement: Synbiotic supplementation — Daily supplementation of synbiotic
  Arms: Synbiotic supplementation; Synbiotic supplementation & dietary intervention
Behavioral: Dietary intervention — Increased fruits and vegetables consumption
  Arms: Dietary intervention; Synbiotic supplementation & dietary intervention

SUMMARY:
Synbiotic is a nutritional supplement that contains both prebiotic and probiotic. Probiotics are beneficial microorganisms, while prebiotics are foods that help the growth of beneficial microorganisms in the gut. In the study, dietary intervention with fruits and vegetables and/or synbiotic supplementation with be administered to Hong Kong Chinese subjects for eight weeks. Changes in the composition and diversity of intestinal microbiota, and markers indicative of obesity, chronic inflammation and metabolic dysfunction will be assessed throughout the whole period. This study will further provide a scientific basis for the intake of synbiotics for reducing the risk of overweight and obesity among Hong Kong Chinese. Furthermore, the results will bridge to further research into the most desirable gut microbiome profile, hence facilitating personalised nutrition for optimal health.

DETAILED DESCRIPTION:
This is an 8-week randomized controlled dietary interventional trial.The objectives of this study include:

* To investigate the effects of synbiotic supplementation and/or dietary intervention with fruits and vegetables on gut microbial diversity and composition, and on inflammation, metabolic functioning, overweight and obesity among Hong Kong Chinese
* To study whether the changes in gut microbial diversity and composition upon the interventions in Hong Kong Chinese are correlated with metabolic functioning and inflammation, as well as overweight or obesity

ELIGIBILITY:
Inclusion Criteria:

* Waist circumference ≥90cm in men and ≥80cm in women
* BMI >23.0kg/m2

Exclusion Criteria:

* Practicing dietary restrictions
* Using cholesterol-lowering, antihypertensive, anti-inflammatory drugs or Chinese medicines
* Consuming laxatives, any gastrointestinal medication, probiotics, prebiotics, synbiotics or antibiotics
* Smokers
* Alcohol abuser
* Currently pregnant or lactating

Ages: 20 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in body weight at week 8 compared with baseline | Week 0, 8
  Body weight in kilogram
Change in Body Mass Index (BMI) at week 8 compared with baseline | Week 0, 8
  BMI = Body weight (in kilograms) divided by square of body height (in meters)
Change in body fat percentage at week 8 compared with baseline | Week 0, 8
  Body fat percentage is assessed by bioimpedence

SECONDARY OUTCOMES:
Change in fasting glucose at week 8 compared with baseline | Week 0, 8
  Fasting glucose in mmol/L
Change in fasting insulin at week 8 compared with baseline | Week 0, 8
  Fasting insulin in pmol/L
Changes in fasting lipids at week 8 compared with baseline | Week 0, 8
  * Triglycerides in mmol/L
  * Total cholesterol in mmol/L
  * HDL-cholesterol in mmol/L
Use of 16S rRNA gene sequencing to assess the changes in the composition of the gut microbiota (bacteriome) of stool samples at week 8 compared with baseline | Week 0, 8
  The composition of the gut microbiota (bacteriome) of stool samples is assessed by 16S rRNA gene sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Hoi Shan Kwan, PhD, Study Chair — Chinese University of Hong Kong; Peter Chi Keung Cheung, PhD, Study Director — Chinese University of Hong Kong; Susana Lauw, MSc, Principal Investigator — Chinese University of Hong Kong; Nelson Kei, BSc, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong